CLINICAL TRIAL: NCT06779877
Title: The Effect of Percutaneous Dilatational Tracheostomy on Intracranial Pressure: a Prospective Observational Study
Brief Title: The Effect of Percutaneous Dilatational Tracheostomy on Intracranial Pressure
Status: Active, not recruiting | Type: Observational
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Melike Cengiz, Professor, Akdeniz University
Other Study IDs: AkdenizU.
Record Dates: First submitted 2025-01-12; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Intracranial Pressure Change; Tracheostomy
Keywords: percutaneous dilatational tracheostomy; optic nerve sheath diameter; intracranial pressure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients without intracranial pathology: Patients undergoing PDT who have been shown to have no intracranial pathology by any imaging procedure
  Interventions: Procedure: Percutaneous dilatational tracheostomy; Diagnostic Test: The optic nerve sheath diameter measurement method by ultrasonography
- Patients with intracranial pathology: Patients undergoing PDT who have been shown to have intracranial pathology by any imaging procedure
  Interventions: Procedure: Percutaneous dilatational tracheostomy; Diagnostic Test: The optic nerve sheath diameter measurement method by ultrasonography

INTERVENTIONS:
Procedure: Percutaneous dilatational tracheostomy — Percutaneous dilatational tracheostomy
Diagnostic Test: The optic nerve sheath diameter measurement method by ultrasonography — The optic nerve sheath diameter measurement method by ultrasonography-Determine intracranial pressure.

SUMMARY:
Percutaneous dilatational tracheostomy (PDT) is a common bedside alternative to surgical tracheostomy in intensive care unit patients. Intracranial pressure measurement is a vital parameter that should be monitored when performing any procedure including PDT in these patients. During PDT, changes in intracranial pressure may occur depending on the position applied, hypercarbia and hypertension that may develop during the procedure. However, the effect of PDT procedure on intracranial pressure is controversial. It is imperative to ascertain the impact of PDT on intracranial pressure, along with the factors that influence its fluctuations during the procedure. This is of particular significance in order to avert the occurrence of deleterious conditions that may be engendered by elevated intracranial pressure. The aim of current study was to evaluate the effect of PDT procedure on intracranial pressure.

DETAILED DESCRIPTION:
Since the study is a prospective observational study, the investigators will not be the decision-making physicians about the treatments applied to the patients. The optic nerve sheath diameter measurement method by ultrasonography will be used to determine intracranial pressure.Intracranial pressure measurement will be performed in neutral position before PDT, after the patient is positioned for the procedure, immediately after the procedure and immediately after the patient is placed in neutral position. Demographic characteristics, comorbidity status, PDT indication, intensive care unit hospitalisation diagnosis, intracranial pathology data, haemodynamic data, arterial blood gas parameters will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Clinical indication for PDT

Exclusion Criteria:

* Age <18
* Patients with glaucoma
* Patients with optic nerve damage
* Patients in whom PDT is contraindicated (coagulopathy, infection at the site of intervention, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 18 who were decided to open percutaneous dilatational tracheostomy for various reasons will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Effect of PDT procedure on intracranial pressure | 6 months
  The primary outcome of this study was to evaluate the impact of bedside PDT on intracranial pressure through ultrasonography-guided measurement of the optic nerve sheath diameter.

SECONDARY OUTCOMES:
The effect of presence/absence of intracranial pathology on intracranial pressure change during PDT procedure | 6 months
  The secondary outcome of this study was to evaluate the effect of the presence/absence of intracranial pathology on intracranial pressure change during bedside PDT procedure by ultrasonography-guided optic nerve sheath diameter measurement.

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)